CLINICAL TRIAL: NCT03873506
Title: Follow-Up Study of Safety and Efficacy of Mesenchymal Stem Cells in Preterm Infants With Moderate or Severe Bronchopulmonary Dysplasia
Brief Title: Follow-Up Study of Mesenchymal Stem Cells for Bronchopulmonary Dysplasia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xia Yunqiu, Director, Children's Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yunqiu xia
Record Dates: First submitted 2019-02-20; First posted 2019-03-13 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; human umbilical cord -derived mesenchymal stem cells
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stem Cell (Experimental): A single intravenous transplantation of Mesenchymal Stem Cell (Dose A - 1 million cells per kg, Dose B - 5 million cells per kg)
  Interventions: Drug: transplantation of hUC-MSCs

INTERVENTIONS:
Drug: transplantation of hUC-MSCs — Human umbilical cord-derived mesenchymal stem cells had given to preterm infants through intravenous infusion.
  Other Names: intravenous infusion of hUC-MSCs

SUMMARY:
This is a follow-up study to investigate the long-term safety and efficacy of human umbilical cord -derived mesenchymal stem cells (hUC-MSCs), for the treatment of BPD in premature infants. Subjects who participated in and completed the initial stage of the PhaseⅠtrial (NCT03558334 ) will be followed-up until 48 months after the hUC-MSCs transplantation.

DETAILED DESCRIPTION:
Subjects who completed the initial stage of the PhaseⅠclinical trial will be followed-up at 5 additional visits: 1, 3, 6, 12 and 24 months after the hUC-MSCs transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who completed the safety and efficacy evaluations in hUC-MSCs PhaseⅠ clinical trial
2. Subject with a written consent form signed by a legal representative or a parent

Exclusion Criteria:

1. Subject whose parent or legal representative does not agree to participate in the study
2. subject who is considered inappropriate to participate the study by the investigator

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Readmission rate | within two years
Duration of the hospital stay due to respiratory infection | within two years

SECONDARY OUTCOMES:
Rate of Survival | within two years
Incidence of Tumorigenicity | within two years
Growth measured by Z-score | within two years
Number of neurological developmental delay | within two years
Number of blindness and deafness | within two years

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Fu, Study Chair — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang YS, Ahn SY, Yoo HS, Sung SI, Choi SJ, Oh WI, Park WS. Mesenchymal stem cells for bronchopulmonary dysplasia: phase 1 dose-escalation clinical trial. J Pediatr. 2014 May;164(5):966-972.e6. doi: 10.1016/j.jpeds.2013.12.011. Epub 2014 Feb 6. PMID 24508444
- [Background] Ahn SY, Chang YS, Kim JH, Sung SI, Park WS. Two-Year Follow-Up Outcomes of Premature Infants Enrolled in the Phase I Trial of Mesenchymal Stem Cells Transplantation for Bronchopulmonary Dysplasia. J Pediatr. 2017 Jun;185:49-54.e2. doi: 10.1016/j.jpeds.2017.02.061. Epub 2017 Mar 21. PMID 28341525